CLINICAL TRIAL: NCT01749098
Title: A Randomized, Subject And Investigator Blinded, Sponsor Open Placebo Controlled, 2 Way, Crossover Phase 1b Study To Examine The Effects Of PF-04958242 On Ketamine Induced Cognitive Impairment In Healthy Male Volunteers
Brief Title: A Study To Examine The Effects Of PF-04958242 On Ketamine-Induced Cognitive Impairment In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1701013
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia
Keywords: PF-04958242; ketamine; cognition; healthy volunteers
MeSH Terms: conditions — Schizophrenia | interventions — PF-04958242; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-04958242 (Experimental): PF-04958242 and ketamine
  Interventions: Drug: PF-04958242; Drug: Ketamine
- Placebo (Placebo Comparator): Placebo and ketamine
  Interventions: Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: PF-04958242 — PF-04958242, 0.35 mg orally administered capsule on Day 1 and 0.25 mg orally administered capsule on Days 2 - 5
  Arms: PF-04958242
Drug: Ketamine — At 60 minutes after the 0.25 mg dose of PF-04958242 on Day 5, Ketamine (0.23 mg/kg over 1 minute, followed by a maintenance rate of 0.58 mg/kg/hr for 75 minutes) will be infused.
  Arms: PF-04958242
Drug: Placebo — Placebo capsule orally administered on Days 1 - 5
  Arms: Placebo
Drug: Ketamine — At 60 minutes after Placebo on Day 5, Ketamine (0.23 mg/kg over 1 minute, followed by a maintenance rate of 0.58 mg/kg/hr for 75 minutes) will be infused.
  Arms: Placebo

SUMMARY:
To assess if PF-04958242 can attenuate the ketamine-induced cognitive impairment in verbal learning and memory, episodic memory and spatial working memory in healthy volunteers.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 21 - 45 years old.
* Able to read and write English as primary language.
* Subjects who are willing to comply with study procedures.

Exclusion Criteria:

* History of any substance abuse or dependence disorder meeting DSM-IV criteria and/or by SCID-NP within the past 12 months, with the exception of nicotine.
* Known sensitivity to ketamine
* Any history of DSM-IV Axis I psychiatric disorders, determined by SCID-NP interview or diagnoses in the view of the investigator.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Test score on the Hopkins Verbal Learning Test - Immediate Recall | Day 5

SECONDARY OUTCOMES:
Test score on the Weschler Digit Span Test | Day 5
Test score on the CogState N-back test | Day 5
Test score on the CogState Spatial Working memory test | Day 5
Test score on the CogState One Card Learning test | Day 5
Test score on the Hopkins Verbal Learning test - Delayed Recall | Day 5
Retrospective rating on the Positive and Negative Syndrome Scale -modified scale' | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, West Haven, Connecticut

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1701013&StudyName=A%20Study%20To%20Examine%20The%20Effects%20Of%20PF-04958242%20On%20Ketamine-Induced%20Cognitive%20Impairment%20In%20Healthy%20Volunteers